CLINICAL TRIAL: NCT01057160
Title: A Study of the Efficacy and Safety of Rizatriptan 10 mg RPD in the Treatment of Acute Migraine in Patients With Non Satisfactory Response to Previous Pharmacologic Treatment
Brief Title: Rizatriptan 10 MG RPD in the Treatment of Acute Migraine
Acronym: Rinotama
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Hans-Christoph Diener, Prof. of Neurology, Universität Duisburg-Essen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MK 462
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- intake of rizatriptan 10 mg (Experimental)
  Interventions: Drug: Rizatriptan
- previous used analgesic (Active Comparator)
  Interventions: Drug: Rizatriptan

INTERVENTIONS:
Drug: Rizatriptan — use of rizatriptan 10 mg for one migraine attack, in comparison to previously used analgetic

SUMMARY:
This is a multicentre, open label, prospective, randomized, two-attack study with active comparator in patients reporting inadequate response to analgesics and/or triptans to examine the efficacy of Rizatriptan 10 mg RPD in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient's signature on the informed consent document [each patient should be given ample time to read (or have read to them) the consent form, ask any questions they may have regarding the trial and have a clear understanding of the trial and the procedures involved prior to the signing of the consent form].
* Have a clinical diagnosis of migraine with or without aura according to IHS criteria at least one year prior to enrollment.
* At screening at least two migraine attacks per month and no more than ten during the last three months prior to inclusion.
* At screening a stable dose of prophylactic medication (including no prophylactic treatment) for at least two months and no change of prophylactic medication during active trial period.

Exclusion Criteria:

* Contraindication to triptans or Rizatriptan according to medical information sheet.
* Patient has a history or clinical evidence of ischemic heart disease (e.g., angina pectoris of any type, history of myocardial infarction or documented silent ischemia) or symptoms or findings consistent with ischemic heart disease, coronary artery vasospasm (including Prinzmetal's variant angina), or other significant underlying cardiovascular disease. Patient has uncontrolled hypertension. Patient has either demonstrated hypersensitivity to or experienced a serious adverse event in response to Rizatriptan or any of its inactive ingredients.
* History of treatment failure for at least one triptan for the treatment of acute migraine attacks.
* Any other headache, except tension type headache on 5 or less days a month within three months prior to screening.
* A history of drug induced headache, medication overuse headache or any other addiction.
* Any history of allergic hypersensitivity or poor tolerance to any components of the preparations used in this trial.
* Females of childbearing potential not using reliable means of birth control, pregnant or lactating females or expected/ planned pregnancy.
* Participation (planned or current) in any investigational drug or device trial within the previous 30 days prior to screening visit.
* Inability to understand the trial procedures, and thus inability to give informed consent.
* History of allergy to sulfa drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2008-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with headache response on a one to four scale after 2 hours. | 2 hours

SECONDARY OUTCOMES:
Percentage of patients being headache free two hours after intake of study medication. Time of dosing to onset of headache relieve. Relief of concomitant symptoms. Rate of sustained pain free Percentage of patients needing rescue medication | (time points 0.5, 1, 1.5, 2, 4, 8, 12, 24 hours after drug intake

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Christoph Diener, Prof., Principal Investigator — Department of Neurology, University Essen
Locations (1):
- Department of Neurology, University Hospital Essen, Essen, Germany